CLINICAL TRIAL: NCT02645188
Title: Effects of Cueing on Gluteus Maximus and Hamstring Recruitment During the Bridging Exercise
Brief Title: Effect of Cueing on Gluteus Maximus Recruitment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John H. Hollman, Ph.D., Professor of Physical Therapy, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-007140
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Muscle Contraction
Keywords: Electromyography; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Cueing
  Interventions: Other: Cueing
- Control (No Intervention)

INTERVENTIONS:
Other: Cueing — Verbal and tactile cueing to enhance gluteus maximus recruitment
  Arms: Experimental

SUMMARY:
Do specific verbal and tactile cues and instructions help people who perform bridging exercises to improve hip muscle strength to optimize recruitment of the gluteus maximus muscle?

ELIGIBILITY:
Inclusion Criteria:

* female
* 18-40 years of age
* normal muscle strength in lower extremities

Exclusion Criteria:

* evidence of patellofemoral pain syndrome
* evidence of femoracetabular impingement
* evidence of mechanical low back pain causing radicular (lower extremity) symptoms
* history of previous hip or knee ligament injury
* history of lower extremity trauma
* history of lower extremity surgery
* history of neurological conditions that impair motor function
* current lower extremity pain that limits functional activities

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Muscle recruitment as a percentage of the maximal voluntary isometric contraction | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Hollman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No